CLINICAL TRIAL: NCT04893928
Title: Role of Information and Communication Technologies for Health Support in Inflammatory Bowel Diseases: The DAMASCO Trial (Stage I)
Brief Title: Role of Information and Communication Technologies for Health Support in Inflammatory Bowel Diseases: The DAMASCO Trial
Acronym: DAMASCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Nacional Profesor Alejandro Posadas (Other)
Collaborators: Hospital Nacional Cayetano Heredia (Unknown); Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: 446 LMiPeS0/21
Record Dates: First submitted 2021-05-07; First posted 2021-05-20 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Inflammatory Bowel Diseases; Knowledge, Attitudes, Practice; Quality of Life; Treatment Adherence and Compliance
Keywords: Social Media; Information and communication technologies
MeSH Terms: conditions — Inflammatory Bowel Diseases; Behavior; Treatment Adherence and Compliance | interventions — Focus Groups; Growth and Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: QUECOMIICAT survey — IBD-related knowledge. It will be assessed using the recently validated QUECOMIICAT (Qüestionari Coneixements Malaltia Inflamatòria Intestinal Catalunya) questionnaire (27) originally developed in Spanish. Compared with the most well-known CCKNOW (Eaden JA et al in 1999)(28), it incorporates IBD updated data (29).
Other: Self-Efficacy for Appropriate Medication Use Scale — Treatment adherence and compliance. It will be assessed using the Self-Efficacy for Appropriate Medication Use Scale (SEAMS), a 13-item self-administered scale previously translated into Spanish and validated by Bozada-Gutiérrez K et al on a Mexican population (3). According to 13 situations asked by the items, patients stratify the level of confidence about correctly taking their medications: 1, not at all confident; 2, somewhat confident; 3, very confident. The sum of results ranges from 13 to 39 points, where higher scores indicate optimal self-efficacy for taking the pharmacological treatment.
Other: ICTs preferences and barriers survey — Information and communication technologies (ICTs) preferences and barriers. It will be assessed using an ad-hoc inventory designed by the authorship. It has 45 questions mainly answered through a 5-points Likert scale. This inventory was inspired by the surveys used by Mauer M et al on an international population with urticaria (11), and those used by Reich J et al (30) and Chowdhary TS et al (31) on American patients with IBD. Survey approaches aspects related to:
  * Frequency of use of ten different ICTs for personal purposes;
  * Frequency of use of ten different ICTs for IBD-related purposes;
  * A free question about others ICTs that the patient uses for IBD-related purposes;
  * Eight specific IBD-related purposes ICTs are used to;
  * Assessment of ICTs for eight IBD-related purposes;
  * Eight Features an IBD-related App must comprehend.
Other: Focus group and IBD mobile App for health support (MAHS) development and validation — In stage II, a qualitative study will be performed using focus group discussion to explore the experiences and perceptions of patients with IBD using ICTs for health support in different contexts. Focus groups will be established following the Krueger and Casey guidelines (32). Collected data will address the development of an IBD MASH. The developed IBD MASH will be validated on a randomised pilot study along stage III. Methodology and ethical aspects of stage II and III will be defined in another proposal, after stage I preliminary findings.

SUMMARY:
In Latin America, inadequate treatment adherence and compliance in IBD patients is around 64% in Brazilians, 54.4% in Mexicans and 50.3% in Argentinians. In industrialised countries, it has been described that in IBD patients, features as younger age, low disease-related knowledge or low treatment adherence and compliance are negatively associated with health-related quality of life (HRQoL). The following research pursues to better understand potential factors related to IBD patients' treatment adherence and compliance as well as patients' IBD-related knowledge level in a Latin American population, and their preferences and barriers when interacting with ICTs for clinical purposes; to develop and to validate an IBD MAHS for Spanish-Speaking patients with Crohn's and ulcerative colitis.

DETAILED DESCRIPTION:
State of the Art:

A chronic condition with a particular approach but also with an unpredictable course difficult treatment adherence and compliance is seen among Inflammatory Bowel Diseases (IBD) patients. In Latin America, inadequate treatment adherence and compliance in IBD patients is around 64% in Brazilians, 54.4% in Mexicans and 50.3% in Argentinians. In the last, a sub-analysis per medication estimated an inadequate adherence in 52.2%, 40.2% and 15.3% for 5-aminosalicylates (5-ASA), thiopurine and biologics, respectively.

In industrialised countries, it has been described that in IBD patients, features as younger age, low disease-related knowledge or low treatment adherence and compliance are negatively associated with health-related quality of life (HRQoL). In Uruguay, IBD annual incidence rate between 2007-2011 was higher in children and young adults (3.45 and 9.12 per 105 habitants) than ≥45 years-old patients (2.92 per 105 habitants). In Chile, using the Crohn's and Colitis Knowledge score (CCKNOW), there were estimated a median score of 9 out of 24 (range 1 - 20). Using the IBD-32 questionnaire in a 50-patients cross-section study, 40% moderate to low HRQoL was identified in Argentina.

Living with chronic diseases is associated with the necessity of self-management education (SME). SME may reduce depression and anxiety, improving HRQoL. As in other chronic diseases, the 90s Internet advent was accompanied by new IBD-related websites, which served mainly as scholarly sources for IBD patients. Since Web 2.0 in the 2000s, social media (including social networks) emergence let users create and share content across digital devices. Web sites, emails, blogs, social media and mobile Applications software (mobile Apps) comprehend Information and communication technologies (ICTs) resources, which facilitates SME through specific disease-related knowledge transfer using the internet.

A United States cross-sectional study demonstrated in 1960 IBD patients that 32% agreed that social media could help disease management. Social media use was higher in IBD younger patients, female, active disease and Crohn's disease. However, 50% could not rate the quality of IBD information posted online, and 68.3% had concerns about privacy or confidentiality. The rising of IBD-related content represented the following limitations: educational content low in quality, non-supervised content by corresponded healthcare providers, and privacy issues.

The popularity of smartphones and tablets has facilitated an increased development of mobile Apps for health support (MAHS) designed by healthcare providers. A good example is the MAHS called myIBDcoach, an HTML web-based tool designed for computers, tablets, and smartphones in the IBD context. Through a randomised trial among Dutch patients, it was demonstrated that a telemedicine intervention with myIBDcoach significantly the baseline treatment adherence improved after a 12-months follow-up (estimated intervention effect of 0.46, 95% IC 0.22 to 0.70; p=0.0002), much more than others health outcomes as HRQoL or disease-related knowledge. Available IBD MAHS consider more clinical care features than mainly education: monitoring, treatment, follow-up, patients' emotions, even bathroom localisation through GPS function.

Problem statement A low disease-related knowledge can influence treatment adherence and compliance in IBD patients, impacting clinical, occupational and social conditions. In the Romanised World, the association between disease-related knowledge and treatment adherence and compliance in IBD patients, or even social issues as work disability, as to how they interact with ICTs for clinical purposes, seems to be more understood in Europe and North America than Latin America. In the last, a better comprehension of these situations is required in order to improve existing treatment adherence and compliance. This context requires more prospective studies in a region with epidemiologic, ethnic and cultural particularities as Latin America, with a rising IBD annual incidence.

An IBD MAHP can play an essential role in reinforcing treatment adherence and compliance in Latin American IBD patients. However, most of the available IBD MAHS is hard-handled, non-validated or non-Spanish language resources. To date, there is only three available in Spanish, but developed in Spain: one in Pediatrics (miEII-PED), and another two addressed to adults patients but still on the validation process (TeleCumple and TECCU). ICTs have demonstrated improved IBD treatment adherence and compliance. Nevertheless, IBD MAHS deserves to be more validated and in the corresponding language and cultural context. We hypothesise that a locally designed, easy-handled IBD MAHS improves IBD-related knowledge and treatment adherence and compliance on IBD patients.

Aims and Scope:

The following research pursues to better understand potential factors related to IBD patients' treatment adherence and compliance as well as patients' IBD-related knowledge level in an Argentinian population, and their preferences and barriers when interacting with ICTs for clinical purposes; to develop and to validate an IBD MAHS for Spanish-Speaking patients with Crohn's and ulcerative colitis.

Materials and methods Study design and settings The DAMASCO trial (Development and Assessment of a Mobile App for Sanitary Support of Spanish-Speaking' with Crohn's and ulcerative Colitis) comprehends three stages. Stage I corresponds to a survey-based prospective cohort observational trial of out-patients in whom IBD-related knowledge level, treatment adherence, compliance, and ICTs preferences and barriers will be assessed in IBD patients. Stage II and III correspond to the design and health outcomes validation of a Spanish-based IBD-MAHP through qualitative study and a randomised trial, respectively.

The DAMASCO trial has been initially conceived as a monocentric study with the participation of IBD patients attended by the Bowel Team, Gastroenterology Service of Hospital Nacional Profesor Alejandro Posadas (HNPAP), El Palomar, Buenos Aires - Argentina, between May 2021 to August 2022. However, the authorship does not discard the future participation of other Argentinian or even from other Latin American Spanish-speaking countries. For the moment, oral confirmation has been obtained from the followings: Instituto Ecuatoriano de Enfermedades Digestivas (IECED, Guayaquil - Ecuador) and Hospital Nacional Cayetano Heredia (HNCH, Lima - Perú). Due to the COVID-19 Pandemic and further worldwide and local politics around the Social Distancing, Quarantine and Isolation, it is foreseen that the study will be started in the second trimester of 2021, during the following two years.

Population Data search strategy. During May 2021, it will be requested to the Department of Statistics and Censuses of each participating centre, records of in-patients and out-patient attention between January 2016 to December 2020 due to the following presumptive or definitive diagnosis following the 10th revision of the International Classification of Diseases (ICD-10): Crohn's disease (ICD-10 K50.0, K50.1, K50.8 and 50.9), ulcerative colitis (ICD-10 K51.0, K51.1, K51.2, K51.3, K51.4, K51.5, K51.8, K51.9), indeterminate colitis or IBD unclassified (ICD-10 K52.3). Selection criteria will be explained below.

Procedure Database recovering and recruitment of patients. A dataset concerning an IBD patients' list attended at each participating centre will be finally performed following selection criteria detailed above, avoiding duplicated cases. For stage I, patients will be recruited by phone or email invitation through the contact information available at corresponding hospital records, but also by personal invitation during Gastroenterology consultation, as long as they belong to the pre-established IBD patients' list. Patients' recruitment will comprehend the acceptance of answering corresponding surveys, which will be available in sheet forms or in an electronic version based on the SurveyMonkey platform. Surveys will comprehend baseline data, IBD-related knowledge, treatment adherence and compliance and ICTs preferences and barriers (explained below).

Focus group and IBD MAHS development and validation. In stage II, a qualitative study will be performed using focus group discussion to explore the experiences and perceptions of patients with IBD using ICTs for health support in different contexts. Focus groups will be established following the Krueger and Casey guidelines. Collected data will address the development of an IBD MASH. The developed IBD MASH will be validated on a randomised pilot study along stage III. Methodology and ethical aspects of stage II and III will be defined in another proposal, after stage I preliminary findings.

Statistical analysis Technical considerations. M.A.P.T. will perform the Statistical Analysis using the latest available R version (R Foundation for Statistical Computing; Vienna, Austria). A p<0.05 will be considered to be statistically significant, but for the univariate-analysis assessment, it will be regarded as a p<0.2, when appropriated.

Sample size. Due to that previously mentioned topics are still pending for larger description among the Latin American population, it is preferred to estimate sample sizes for exploratory analysis. The total number of patients registered in the prospective IBD database of a digestive centre in La Argentina (n=4000) has been considered as a reference for the universe. It has been decided a margin of error of 5% and a confidence interval (CI) of 95%. Proportions estimation considers finite population correction, and it has been calculated using the R function sample.size.prop.

* Considering that around 29% of Chilean IBD patients answered correctly more than 50% of CCKNOW, the sample size for estimating this IBD-related knowledge level rate on our population will be n=294.
* Considering that around 50.3% of Argentinian IBD patients have inadequate treatment adherence, the sample size for estimating the rate of treatment adherence and compliance in our population will be n=351.
* Considering that around 16.7% of American IBD patients use social media to obtain or post IBD-related information, the sample size for estimating this aspect on our population will be n=203.

Descriptive analysis. Quantitative variables will be described in means (standard deviation, SD) or median (minimum-maximum range) following statistical distribution (Kolmogórov-Smirnov test). Qualitative variables will be described in frequency (%), and the 95% CI will be calculated when necessary.

Inferential analysis:

* Psychometrical testing of QUECOMIICAT: Cronbach's alpha coefficient, principal component analysis (PCA), test-retest reliability.
* Association between QUECOMIICAT and SEAMS: linear regression.
* Risk factors modelling: univariate and multivariate are based on logistic regression (OR, Odds Ratio).

Ethics The DAMASCO trial (stage I) has been approved by the Institutional Review Board (IRB) of the HNPAP. In order to use the previously mentioned surveys, the authorship has obtained corresponding authorisation from the authors of QUECOMIICAT questionary, Spanish-validated version of SEAMS, and surveys which inspired designed ICTs preferences and barriers instrument used on this research. Enrolled patients will sign an informed consent before answering respective surveys along stage I. A brief study explanation will be attached to the surveys. Stage II and III ethic aspects will be discussed after stage I preliminary findings and detailed in a subsequent research proposal. Patient identity and record confidentiality will be granted as described by Law Nº 25.326 Personal Data Protection (Ministry of Justice and Human Rights, Argentine Republic). The study will be conducted in adherence to the 1947 Nuremberg Code and the 1964 Declaration of Helsinki, and later amendments (the latest in 2013).

ELIGIBILITY:
Inclusion Criteria:

* Every patient ≥15 years old;
* Patients attended by a Gastroenterology consultation;
* Patients attended due to an established diagnosis of Crohn's disease, ulcerative colitis, indeterminate colitis or IBD unclassified;
* Patients whose diagnosis should be based on Lennard-Jonnes criteria: clinical, imaging, endoscopic or anatomopathological findings.

Exclusion Criteria:

* Patients with a recent diagnosis and no more than a 6-months follow-up;
* Patients ongoing hospitalisation due to severe IBD flare;
* Patients with psychiatric diseases, language impairment, those who find it difficult to visualise the survey or any other condition that difficult answering of a self-administered survey;
* Patients who they are sanitary professional will not be considered for disease-related knowledge level evaluation;
* Patients not under pharmacological treatment (as naïve patients) will not be considered for treatment adherence and compliance evaluation

Ages: 15 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Out-patients with IBD confirmed diagnosis, to who they are attended at one of the centres participating in this study.
Sampling Method: Non-Probability Sample
Enrollment: 351 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
IBD-related knowledge level | One year
  IBD-related knowledge will be assessed using the recently validated QUECOMIICAT (Qüestionari Coneixements Malaltia Inflamatòria Intestinal Catalunya) questionnaire, originally developed in Spanish. Compared with the most well-known CCKNOW, it incorporates IBD updated data. The QUECOMIICAT questionnaire has 25 multiple-choice questions with four options and only one correct answer. Final questionnaire score ranges from 0 to 25.
Treatment adherence and compliance | One year
  It will be assessed using the Self-Efficacy for Appropriate Medication Use Scale (SEAMS), a 13-item self-administered scale previously translated and validated to Spanish. Along 13 questions, patients stratify the level of confidence about correctly taking their medications:
  1. Not at all confident (1 point);
  2. Somewhat confident (2 points);
  3. Very confident (3 points).
  The sum of results will range from 13 to 39 points. A score 39/39 will be interpreted as the optimal self-efficacy for taking the pharmacological treatment, and a score of 13/39, the lowest.
Information and communication technologies preferences and barriers | One year
  It will be assessed using an ad-hoc inventory designed by the authorship. It has 45 questions mainly answered through a 5-points Likert scale. Survey approaches aspects related to:
  1. Frequency of use of ten different ICTs for personal purposes;
  2. Frequency of use of ten different ICTs for IBD-related purposes;
  3. A free question about other ICTs that the patient uses for IBD-related purposes;
  4. Eight specific IBD-related purposes ICTs are used to;
  5. Assessment of ICTs for eight IBD-related purposes;
  6. Eight Features an IBD-related App must comprehend.
  The 18 questions from point b and d will be useful for estimating how much do IBD patients use ICTs for IBD purposes. Questions will be scored from 1 (never or completely disagree) to 5 (daily use or completely agree). A final score will be summarized from 18 to 90. A score of 18/90 will mean the lowest frequency of ICTs use for IBD purposes, and 90/90 the highest.

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Angel Puga Tejada, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoivik ML, Moum B, Solberg IC, Henriksen M, Cvancarova M, Bernklev T; IBSEN Group. Work disability in inflammatory bowel disease patients 10 years after disease onset: results from the IBSEN Study. Gut. 2013 Mar;62(3):368-75. doi: 10.1136/gutjnl-2012-302311. Epub 2012 Jun 20. PMID 22717453
- [Background] Cornelio Rde C, Pinto AL, Pace FH, Moraes JP, Chebli JM. [Non-adherence to the therapy in Crohn's disease patients: prevalence and risk factors]. Arq Gastroenterol. 2009 Jul-Sep;46(3):183-9. doi: 10.1590/s0004-28032009000300008. Portuguese. PMID 19918683
- [Background] Bozada-Gutierrez KE, Fresan-Orellana A, Yamamoto-Furusho JK. Validacion de Belief Medicines Questionnaire y Self-efficacy for Appropriate Medication Use Scale para medir adherencia al tratamiento farmacologico en pacientes con enfermedad inflamatoria intestinal. Gac Med Mex. 2019;155(2):124-129. doi: 10.24875/GMM.18004417. PMID 31056588
- [Background] Lasa J, Correa G, Fuxman C, Garbi L, Linares ME, Lubrano P, Rausch A, Toro M, Yantorno M, Zubiaurre I, Peyrin-Biroulet L, Olivera P. Treatment Adherence in Inflammatory Bowel Disease Patients from Argentina: A Multicenter Study. Gastroenterol Res Pract. 2020 Jan 17;2020:4060648. doi: 10.1155/2020/4060648. eCollection 2020. PMID 32411197
- [Background] Gomollon F. Treatment adherence is always worse than we think: an unresolved problem in inflammatory bowel disease. Gastroenterol Hepatol. 2016 Sep;39 Suppl 1:14-19. doi: 10.1016/S0210-5705(16)30170-4. English, Spanish. PMID 27888859
- [Background] Leong RW, Lawrance IC, Ching JY, Cheung CM, Fung SS, Ho JN, Philpott J, Wallace AR, Sung JJ. Knowledge, quality of life, and use of complementary and alternative medicine and therapies in inflammatory bowel disease: a comparison of Chinese and Caucasian patients. Dig Dis Sci. 2004 Oct;49(10):1672-6. doi: 10.1023/b:ddas.0000043384.26092.f4. PMID 15573925
- [Background] Hommel KA, Davis CM, Baldassano RN. Medication adherence and quality of life in pediatric inflammatory bowel disease. J Pediatr Psychol. 2008 Sep;33(8):867-74. doi: 10.1093/jpepsy/jsn022. Epub 2008 Mar 11. PMID 18337262
- [Background] Simian D, Flores L, Quera R, Kronberg U, Ibanez P, Figueroa C, Lubascher J. Assessment of disease-related knowledge and possible factors associated with the knowledge level among Chilean patients with inflammatory bowel disease. J Clin Nurs. 2017 Jun;26(11-12):1508-1515. doi: 10.1111/jocn.13436. Epub 2017 Mar 20. PMID 27322103
- [Background] Rodríguez-Núñez MG, Conlon MC, Spiazzi RA, Canicoba M, Milano MC. Evaluar la calidad de vida en pacientes con enfermedad inflamatoria intestinal mediante el cuestionario IBDQ-32. Acta Gastroenterol Latinoam. 2016;46(S1):2016.
- [Background] Vettorato MG, Lorenzon G, Marchi E De, Ottavia Bartolo F, Cavallin R, Rigo A, et al. Mo1859 Patient Support Programme Is Well Accepted And Could Help Adherence In IBD Patients. Gastroenterology [Internet]. 2016;150(4):S797. Available from: http://dx.doi.org/10.1016/S0016-5085(16)32702-0
- [Background] Maurer M, Weller K, Magerl M, Maurer RR, Vanegas E, Felix M, Cherrez A, Mata VL, Kasperska-Zajac A, Sikora A, Fomina D, Kovalkova E, Godse K, Rao ND, Khoshkhui M, Rastgoo S, Criado RFJ, Abuzakouk M, Grandon D, van Doorn M, Valle SOR, de Souza Lima EM, Thomsen SF, Ramon GD, Matos Benavides EE, Bauer A, Gimenez-Arnau AM, Kocaturk E, Guillet C, Ignacio Larco J, Zhao ZT, Makris M, Ritchie C, Xepapadaki P, Ensina LF, Cherrez S, Cherrez-Ojeda I. The usage, quality and relevance of information and communications technologies in patients with chronic urticaria: A UCARE study. World Allergy Organ J. 2020 Oct 30;13(11):100475. doi: 10.1016/j.waojou.2020.100475. eCollection 2020 Nov. PMID 33204387
- [Background] Soetikno RM, Provenzale D, Lenert LA. Studying ulcerative colitis over the World Wide Web. Am J Gastroenterol. 1997 Mar;92(3):457-60. PMID 9068469
- [Background] Kaplan AM. If you love something, let it go mobile: Mobile marketing and mobile social media 4x4. Bus Horiz [Internet]. 2012;55(2):129-39. Available from: http://dx.doi.org/10.1016/j.bushor.2011.10.009
- [Background] Reich J, Guo L, Groshek J, Weinberg J, Chen W, Martin C, Long MD, Farraye FA. Social Media Use and Preferences in Patients With Inflammatory Bowel Disease. Inflamm Bowel Dis. 2019 Feb 21;25(3):587-591. doi: 10.1093/ibd/izy280. PMID 30203036
- [Background] Mukewar S, Mani P, Wu X, Lopez R, Shen B. YouTube and inflammatory bowel disease. J Crohns Colitis. 2013 Jun;7(5):392-402. doi: 10.1016/j.crohns.2012.07.011. Epub 2012 Aug 18. PMID 22906403
- [Background] Fortinsky KJ, Fournier MR, Benchimol EI. Internet and electronic resources for inflammatory bowel disease: a primer for providers and patients. Inflamm Bowel Dis. 2012 Jun;18(6):1156-63. doi: 10.1002/ibd.22834. Epub 2011 Dec 6. PMID 22147497
- [Background] de Jong MJ, van der Meulen-de Jong AE, Romberg-Camps MJ, Becx MC, Maljaars JP, Cilissen M, van Bodegraven AA, Mahmmod N, Markus T, Hameeteman WM, Dijkstra G, Masclee AA, Boonen A, Winkens B, van Tubergen A, Jonkers DM, Pierik MJ. Telemedicine for management of inflammatory bowel disease (myIBDcoach): a pragmatic, multicentre, randomised controlled trial. Lancet. 2017 Sep 2;390(10098):959-968. doi: 10.1016/S0140-6736(17)31327-2. Epub 2017 Jul 14. PMID 28716313
- [Background] Yin AL, Hachuel D, Pollak JP, Scherl EJ, Estrin D. Digital Health Apps in the Clinical Care of Inflammatory Bowel Disease: Scoping Review. J Med Internet Res. 2019 Aug 19;21(8):e14630. doi: 10.2196/14630. PMID 31429410
- [Background] Calderon M, Minckas N, Nunez S, Ciapponi A. Inflammatory Bowel Disease in Latin America: A Systematic Review. Value Health Reg Issues. 2018 Dec;17:126-134. doi: 10.1016/j.vhri.2018.03.010. Epub 2018 Jun 22. PMID 29936359
- [Background] Cerezo MJ, Conlon MC, Milano MC, Spiazzi RA. Parasitosis en enfermedad inflamatoria intestinal. Acta Gastroenterol Latinoam. 2019;46:S9.
- [Background] Yamamoto-Furusho JK, Bosques-Padilla FJ, Charua-Guindic L, Cortes-Espinosa T, Miranda-Cordero RM, Saez A, Ledesma-Osorio Y. Inflammatory bowel disease in Mexico: Epidemiology, burden of disease, and treatment trends. Rev Gastroenterol Mex (Engl Ed). 2020 Jul-Sep;85(3):246-256. doi: 10.1016/j.rgmx.2019.07.008. Epub 2020 Mar 3. English, Spanish. PMID 32143974
- [Background] Del Hoyo JD, Nos P, Faubel R, Bastida G, Munoz D, Valero-Perez E, Garrido-Marin A, Bella P, Pena B, Savini C, Aguas M. Adaptation of TECCU App Based on Patients Perceptions for the Telemonitoring of Inflammatory Bowel Disease: A Qualitative Study Using Focus Groups. Int J Environ Res Public Health. 2020 Mar 13;17(6):1871. doi: 10.3390/ijerph17061871. PMID 32183103
- [Background] Pedersen N, Thielsen P, Martinsen L, Bennedsen M, Haaber A, Langholz E, Vegh Z, Duricova D, Jess T, Bell S, Burisch J, Munkholm P. eHealth: individualization of mesalazine treatment through a self-managed web-based solution in mild-to-moderate ulcerative colitis. Inflamm Bowel Dis. 2014 Dec;20(12):2276-85. doi: 10.1097/MIB.0000000000000199. PMID 25248002
- [Background] Cross RK, Jambaulikar G, Langenberg P, Tracy JK, Collins JF, Katz J, Regueiro M, Schwartz DA, Quinn CC. TELEmedicine for Patients with Inflammatory Bowel Disease (TELE-IBD): Design and implementation of randomized clinical trial. Contemp Clin Trials. 2015 May;42:132-44. doi: 10.1016/j.cct.2015.03.006. Epub 2015 Mar 24. PMID 25812483
- [Background] Presidencia de la Nación. Distanciamiento social, preventivo y obligatorio (DISPO) y aislamiento social, preventivo y obligatorio (ASPO). Boletín Of la República Argentina. 2021;125.
- [Background] Lennard-Jones J. Crohn's disease: definition, pathogenesis, aetiology. Clin Gastroenterol. 1980;173-89.
- [Background] Casellas F, Navarro E, Amil P, Barber C, Marin L, Guardiola J, Espin E, Sainz E, Aldeguer X, Gallego M, Murciano F, Garcia-Planella E, Martin-de-Carpi J, Mendive JM, Gonzalez-Mestre A. Development and validation of the QUECOMIICAT questionnaire: a tool to assess disease-related knowledge in patients with inflammatory bowel disease. Rev Esp Enferm Dig. 2019 Aug;111(8):586-592. doi: 10.17235/reed.2019.6298/2019. PMID 31317762
- [Background] Eaden JA, Abrams K, Mayberry JF. The Crohn's and Colitis Knowledge Score: a test for measuring patient knowledge in inflammatory bowel disease. Am J Gastroenterol. 1999 Dec;94(12):3560-6. doi: 10.1111/j.1572-0241.1999.01536.x. PMID 10606319
- [Background] Yoon H, Yang SK, So H, Lee KE, Park SH, Jung SA, Choh JH, Shin CM, Park YS, Kim N, Lee DH. Development, validation, and application of a novel tool to measure disease-related knowledge in patients with inflammatory bowel disease. Korean J Intern Med. 2019 Jan;34(1):81-89. doi: 10.3904/kjim.2017.104. Epub 2017 Nov 29. PMID 29172400
- [Background] Chowdhary TS, Thompson J, Gayam S. Social Media Use for Inflammatory Bowel Disease in a Rural Appalachian Population. Telemed J E Health. 2021 Apr;27(4):402-408. doi: 10.1089/tmj.2020.0014. Epub 2020 Jun 18. PMID 32552561
- [Background] Krueger R, Casey M. Focus Groups: A Practical Guide for Applied Research,. 5th ed. CA, USA: SAGE Publications Inc.; 2015.
- [Background] Sambuelli AM, Toro MA, Negreira SM, Gil AH, Goncalves SA, Huernos SP, Bai JC. [Activity index in Crohn's disease]. Acta Gastroenterol Latinoam. 2005;35(1):28-36. Spanish. PMID 15954734
- [Background] Chow S, Shao J, Wang H. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series, editor. 2008. 89 p.
- [Background] Kauermann G, Kuechenhoff H. Stichproben. Methoden und praktische Umsetzung mit R. Springer; 2010.
- [Background] Ruíz-Morales Á, Gómez-Restrepo C. Epidemiología Clínica: investigación clínica aplicada. Editorial Médica Panamericana; 2015.
- [Background] Ventura-León J. Educación Médica. Educ Médica. 2020;21(3):218-20.